CLINICAL TRIAL: NCT02906189
Title: Safety of Magnetic Resonance Imaging in Non-MRI Conditional Pacemakers and ICD Devices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Banner Health (Other)
Responsible Party: Principal Investigator, Michael Morris, Clinical Assistant Professor, Banner Health
Other Study IDs: 1608820677
Record Dates: First submitted 2016-09-03; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: MRI

SUMMARY:
The primary objective of the study is to determine the safety of MRI in patients with non-MRI conditional pacemakers. The secondary objective is to determine if there are clinically relevant parameter changes in the devices.

ELIGIBILITY:
Inclusion Criteria. All patients with non-MRI conditional pacemakers and ICDs between the ages of 18-85 will be eligible to participate. Medical records will be reviewed to confirm the date and make/model of device implanted. Ordering physician discusses the MRI request with radiologist, documenting that there is no appropriate alternate imaging test. Patient must have an appointment with a cardiologist/electrophysiologist prior to MRI. Banner Health policy for standard of care guidelines involving patients receiving MRI's will be followed.

Exclusion Criteria. Patients will be excluded from MRI based on the Department of Radiology protocol. Additional exclusion criteria include: ICD and pacemaker dependent, Pacemaker inserted before 2002, Epicardial leads, fractured leads, abandoned leads, or temporary pacemakers (post-coronary artery bypass graft temporary epicardial pacing wires are acceptable), Patient not awake or unable communicate, Battery voltage at elective replacement interval, implanted non-MRI conditional device (other than pacemaker/ICD).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-MRI conditional pacemakers and ICDs referred for clinically indicated MRI scans.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Death during the MRI scan | Immediate

SECONDARY OUTCOMES:
Decrease in battery voltage >0.04v | 6 months
Change in pacing lead impedance ≥ 50 Ω | 6 months
Change in high-voltage lead impedance ≥ 3 Ω | 6 months
Increase in pacing threshold ≥ 0.50 V @ 0.4 ms | 6 months
Decrease in P wave measurement ≥ 50% | 6 months
Decrease in R wave measurement ≥ 25% | 6 months
Generator failure requiring immediate replacement | Immediate
Lead failure requiring immediate replacement | Immediate
New onset atrial or ventricular arrhythmia during MRI | Immediate
Loss of pacemaker capture during MRI | Immediate
Electrical reset of the device | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Banner University Medical Center
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No